CLINICAL TRIAL: NCT05282745
Title: A Multicenter Cohort Study of HPV Viral Load in Predicting the Postoperative Recurrence of Women With HSIL in Cervix
Brief Title: A Multicenter Cohort Study of HPV Viral Load in Predicting the Postoperative Recurrence of HSIL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fujian Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, Binhua Dong, Principal Investigator, Fujian Maternity and Child Health Hospital
Other Study IDs: PVLHCF
Record Dates: First submitted 2022-02-17; First posted 2022-03-16 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: HPV Infection; HSIL, High-Grade Squamous Intraepithelial Lesions; Viral Load
MeSH Terms: conditions — Papillomavirus Infections; Squamous Intraepithelial Lesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — DNA samples from cervix and vaginal fornix & cell samples from cervix
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with high-grade squamous intraepithelial lesion (HSIL) in cervix: In the enrollment, women whose cervical histopathological results have been diagnosed as high-grade squamous intraepithelial lesion (HSIL) for the last 3 months with abnormal results will be included in this study. All participants will be followed up three times, at 6 months,12 months and 24 months.
  Interventions: Other: Follow-up

INTERVENTIONS:
Other: Follow-up — Participants will be followed up at 6, 12 and 24 months with HPV viral load tests, Thinprep cytologic tests (TCT) and vaginal secretion tests.

SUMMARY:
Human papillomavirus (HPV) infection has become one of the most important health problems faced by women all over the world. A large number of studies have shown that women's cervical, vaginal and perianal precancerous lesions, related cancers, condyloma acuminatum and other sexually transmitted diseases (STD) are closely related to HPV infection. Among them, the persistent infection of high-risk human papillomavirus (HR-HPV) is closely related to the occurrence of invasive cervical cancer. Previous studies have shown that there are significant differences in the effects of multiple HPV infection and persistent infection of different types (such as type-16, -18, -39 and -52) on different levels of cervical lesions, and there is a certain correlation between HPV load in the process of persistent infection and the degree of cervical lesions. In addition, other studies have shown that HPV-16 viral load has certain clinical significance in predicting Cin2 / CIN3 high-grade cervical lesions, and HPV viral load level is significantly different in cervical low-grade squamous intraepithelial lesion (LSIL) and cervical high-grade squamous intraepithelial lesion (HSIL). The above biological changes such as HPV infection type, quantity and proportion can promote the occurrence and development of cervical precancerous lesions and related cancers to varying degrees. It can be seen that the study of the relationship between HPV viral load and cervical lesions is of great significance for clinical disease development prediction and cervical cancer screening.

DETAILED DESCRIPTION:
Based on previous studies and clinical practice, this study carried out a multi center cohort study in China. In this study, ten research including Fujian Maternity and Child Health Hospital, Mindong Hospital of Ningde City, Zhangzhou affiliated Hospital of Fujian Medical University, Quanzhou First Hospital Afflicated to Fujian Medical University, The First Hospital of Putian City, Ningde Municipal Hospital of Ningde Normal University, Shenzhen Maternity and child Healthcare Hospital and Maternity and child Hospital of Hubei Province were included, each of which included 400 individuals, with a total of 4000 women with high-grade squamous intraepithelial lesion were enrolled. For the first time, the investigators will collect 2 samples of cervical exfoliated cells and 4 samples of vaginal fornix swabs from participants, then at the 6th, 12th and 24th months after the first sampling, the participants need to return to the hospital, collected 2 samples of cervical exfoliated cells and 4 samples of vaginal fornix swabs again in order to observe and record the development of the disease. During this process, if abnormal cervical lesions are found, the participants will be biopsied under colposcopy according to relevant guidelines. Samples from cervix would be sent for PCR-sequencing, HPV tests and Thinprep cytologic test (TCT). And samples from vaginal fornix would be sent for sequencing and bioinformatic analysis. A prospective cohort study was conducted to explore the correlation between the characteristics, progression and prognosis of female genital tract lesions and HPV infection type, load and vaginal microenvironment.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20 and over.
* The result of cervical histopathology in the last 3 months was high-grade squamous intraepithelial lesion (HSIL).
* Non pregnant people with sexual history.
* Asexual life, no vaginal medication or flushing before 72 hours of sampling.

Exclusion Criteria:

* Within 8 weeks after pregnancy or postpartum.
* Patients with history of genital tract tumor.
* History of HPV vaccination.
* Previous history of hysterectomy, cervical surgery, pelvic radiotherapy Historical.
* In recent one month, she has received genital tract infection, HPV or other STDs treatment related to the infection of mycoplasma.
* Use antibiotics or vaginal microecological improvement products in recent 1 month.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese women aged 20 and over with high-grade squamous intraepithelial lesion in results of cervical histopathology.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Cervical histopathology testing at baseline | Baseline
  Cervical histopathology was performed at baseline for all participants.
Cervical histopathology testing at 6-month follow-up | 6-month follow-up
  Cervical histopathology was performed at 6-month follow-up for cervical HPV infection or cytology abnormalities women.
Cervical histopathology testing at 12-month follow-up | 12-month follow-up
  Cervical histopathology was performed at 12-month follow-up for cervical HPV infection or cytology abnormalities women.
Cervical histopathology testing at 24-month follow-up | 24-month follow-up
  Cervical histopathology was performed at 24-month follow-up for cervical HPV infection or cytology abnormalities women.
Human Papillomavirus (HPV) viral load test at baseline | Baseline
  Human Papillomavirus (HPV) viral load test was performed at baseline for all participants.
Human Papillomavirus (HPV) viral load test at 6-month follow-up | 6-month follow-up
  All participants were tested for HPV viral load at the time of 6-month follow-up.
Human Papillomavirus (HPV) viral load test at 12-month follow-up | 12-month follow-up
  All participants were tested for HPV viral load at the time of 12-month follow-up.
Human Papillomavirus (HPV) viral load test at 24-month follow-up | 24-month follow-up
  All participants were tested for HPV viral load at the time of 24-month follow-up.
Cervical cytology testing at baseline | Baseline
  All participants were tested for cervical cytology at the time of baseline.
Cervical cytology testing at 6-month follow-up | 6-month follow-up
  All participants were tested for Cervical cytology testing at the time of 6-month follow-up.
Cervical cytology testing at 12-month follow-up | 12-month follow-up
  All participants were tested for Cervical cytology testing at the time of 12-month follow-up.
Cervical cytology testing at 24-month follow-up | 24-month follow-up
  All participants were tested for Cervical cytology testing at the time of 24-month follow-up.
16SrRNA sequencing of the vaginal secretions at baseline | Baseline
  All participants underwent vaginal secretion sequencing at baseline.
16SrRNA sequencing the vaginal secretions at 6-month follow-up | 6-month follow-up
  All participants underwent vaginal secretion sequencing at the time of 6-month follow-up.
16SrRNA sequencing of the vaginal secretions at 12-month follow-up | 12-month follow-up
  All participants underwent vaginal secretion sequencing at the time of 12-month follow-up.
16SrRNA sequencing of the vaginal secretions at 24-month follow-up | 24-month follow-up
  All participants underwent vaginal secretion sequencing at the time of 24-month follow-up.

SECONDARY OUTCOMES:
Human Papillomavirus (HPV) genotyping tests at baseline | Baseline
  All participants underwent Human Papillomavirus (HPV) genotyping tests at baseline.
Human Papillomavirus (HPV) genotyping tests at 6-month follow-up | 6-month follow-up
  All participants underwent Human Papillomavirus (HPV) genotyping tests at the time of 6-month follow-up.
Human Papillomavirus (HPV) genotyping tests at 12-month follow-up | 12-month follow-up
  All participants underwent Human Papillomavirus (HPV) genotyping tests at the time of 12-month follow-up.
Human Papillomavirus (HPV) genotyping tests at 24-month follow-up | 24-month follow-up
  All participants underwent Human Papillomavirus (HPV) genotyping tests at the time of 24-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Pengming Sun, PhD, Study Chair — Fujian Maternity and Child Health Hospital, Affiliated Hospital of Fujian Medical University
Locations (10):
- China (10):
  - Fujian Maternity and Child Health Hospital, Fuzhou, Fujian
  - Mindong Hospital of Ningde City, Ningde, Fujian
  - Ningde Municipal Hospital of Ningde Normal University, Ningde, Fujian
  - The First Hospital of Putian City, Putian, Fujian
  - Quanzhou First Hospital Afflicated to Fujian Medical University, Quanzhou, Fujian
  - Zhangzhou affiliated Hospital of Fujian Medical University, Zhangzhou, Fujian
  - Longyan First Hospital, Longyan
  - Shenzhen Maternity and child Healthcare Hospital, Shenzhen
  - Maternity and child Hospital of Hubei Province, Wuhan
  - Xiamen Maternity and Child Health Hospital, Xiamen